CLINICAL TRIAL: NCT05559281
Title: Evaluation of Botulinum Toxin Injection in Reducing Lip Scar Following Cleft Lip Repair (Randomized Controlled Clinical Trial)
Brief Title: Botulinum Toxin Injection in Reducing Lip Scar Following Cleft Lip Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Botulinum_2020
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Cleft Lip
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Botulinum
- Group B (Active Comparator)
  Interventions: Procedure: Fisher technique

INTERVENTIONS:
Other: Botulinum — injection of Botulinum Toxin injection in lip muscles following cleft lip repair surgically.
  Arms: Group A
Procedure: Fisher technique — The cleft lip will be treated surgically using the Fisher technique only.
  Arms: Group B

SUMMARY:
A cleft lip is a congenital defect resulting from failing to merge developmental processes in the Orofacial region. One of the most common complications surgeons fear after cleft lip repair is a hypertrophic scar. A cleft scar negatively affects a patient's appearance, psychology, and function. Several techniques have been proposed to improve lip scars such as steroid therapy, laser therapy, and silica gel. Despite such efforts, the results were still unsatisfactory. Botulinum Toxin injections may provide a more reliable method

ELIGIBILITY:
Inclusion Criteria:

* With mild to severe cleft lip deformity requiring repair.
* Neonates up to 1 year of age.
* Patients with or without cleft palate.
* Systemically healthy patients.
* Patients follow postoperative instructions provided by their legal guardians.

Exclusion Criteria:

* Patients with a syndromic type of cleft lip.
* Patients suffering from relevant systemic and metabolic diseases.
* Patients suffering from immunosuppressive diseases.
* Patients suffering from neuromuscular disorders like Myasthenia Gravis.
* Patients with special needs.

Ages: 0 Minutes to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in cleft scar | 2 weeks, 3 months, 6 months
  Vancouver Scar Scale: This scale focuses on four parameters:
  scar height and thickness, pliability, vascularity, and pigmentation to generate a score ranging from 0 to 13 point

SECONDARY OUTCOMES:
Change in scar width | 2 weeks, 3 months, 6 months
  The scar width is to be measured at two certain points using digital caliper, one point is 1 mm above white line and the second point is 1 mm below nasal
Change in lip height | 2 weeks, 3 months, 6 months
  The lip height measurement will be done using digital caliper at cleft and non-cleft side.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt